CLINICAL TRIAL: NCT07147036
Title: Comparison of Effectiveness of Biodentine Versus Calcium Hydroxide as Indirect Pulp Capping Material in Mature Permanent Teeth
Brief Title: Effectiveness of Biodentine v/s Calcium Hydroxide as Indirect Pulp Capping Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahoor khan (Other)
Collaborators: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Zahoor khan, Dr Zahoor khan, Resident operative dentistry & endodontics, HITECIMS taxila pakistan, HITEC-Institute of Medical Sciences
Organization: HITEC-Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dental/HITEC/IRB/41
Record Dates: First submitted 2025-08-08; First posted 2025-08-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Reversible Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biodentine Group (Experimental): Participants receive Biodentine as the indirect pulp capping material
  Interventions: Procedure: Biodentine - Indirect Pulp Capping
- Calcium Hydroxide Group (Active Comparator): Participants receive Calcium Hydroxide (Dycal) as the indirect pulp capping material
  Interventions: Procedure: Calcium Hydroxide - Indirect Pulp Capping

INTERVENTIONS:
Procedure: Biodentine - Indirect Pulp Capping — Caries removal under rubber dam isolation using round bur (#BR-45) and water spray
  Tooth disinfection with 0.2% chlorhexidine
  Mixing of Biodentine (Septodont, France) in an amalgamator (30 seconds at 4000 rpm)
  Placement of Biodentine into the prepared cavity using an amalgam carrier and condensation
  After 1 week: Placement of self-cure GIC (Fuji, Japan) as a base
  Final restoration with light-cure composite resin
  Follow-up at 2, 6, and 12 weeks
  Arms: Biodentine Group
Procedure: Calcium Hydroxide - Indirect Pulp Capping — Caries removal under rubber dam isolation using round bur (#BR-45) and water spray
  Tooth disinfection with 0.2% chlorhexidine
  Cavity dried with cotton pellet
  Placement of a 0.5 mm layer of Calcium Hydroxide (Dycal)
  After 2-3 minutes (setting time): Placement of self-cure GIC (Fuji, Japan)
  After 1 week: Final restoration with light-cure composite resin
  Follow-up at 2, 6, and 12 weeks
  Arms: Calcium Hydroxide Group

SUMMARY:
This study compares the clinical and radiographic effectiveness of Biodentine and Calcium Hydroxide as indirect pulp capping materials in mature permanent teeth with reversible pulpitis. A total of 76 patients were randomly assigned to two groups. Outcomes were assessed over 12 weeks based on pain, periapical radiolucency, and PDL widening. The goal was to determine which material better preserves pulp vitality

DETAILED DESCRIPTION:
Introduction:

Preservation of pulp vitality is critical for the long-term health and functionality of teeth. The pulp can be compromised due to caries, trauma, or iatrogenic factors. One conservative treatment to preserve pulp vitality in teeth with deep carious lesions and reversible pulpitis is indirect pulp capping (IPC).

Traditionally, Calcium Hydroxide (Ca(OH)₂) has been the gold standard material for IPC due to its antibacterial properties and its ability to stimulate the formation of reparative dentin. However, it has several limitations such as poor bonding to dentin, high solubility, and low mechanical strength, which may affect long-term success.

Biodentine, a newer bioactive dentin substitute, has emerged as a potential alternative due to its biocompatibility, bioactivity, antibacterial effect, good sealing ability, and high compressive strength. These properties suggest Biodentine may offer superior clinical outcomes in preserving pulp vitality when used as an indirect pulp capping material.

Objective:

To compare the clinical and radiographic effectiveness of Biodentine versus Calcium Hydroxide as indirect pulp capping agents in mature permanent teeth with reversible pulpitis.

Study Design:

Type: Experimental comparative study

Setting: Department of Operative Dentistry & Endodontics, HITEC-IMS, Taxila

Duration: 1 year (after IRB approval)

Sample Size: 76 patients (38 in each group), calculated using WHO sample size calculator

Sampling Technique: Non-probability consecutive sampling

Inclusion Criteria:

Patients aged 20-45 years

Teeth with occlusal carious lesions with ICDAS radiographic score RC-5

Vital teeth with signs of reversible pulpitis

No signs of root resorption

Exclusion Criteria:

Teeth tender to percussion

Irreversible pulpitis or non-vital pulp

Medically compromised or pregnant patients

Third molars or teeth with pulp exposure during caries excavation

Materials Used:

Group I: Biodentine (Septodont, France)

Group II: Calcium Hydroxide (Dycal)

Base Material: Self-cure Glass Ionomer Cement (Fuji, Japan)

Final Restoration: Light-cure composite resin

Disinfectant: 0.2% Chlorhexidine

Vitality Tests: Cold test and electric pulp test

Caries Removal: Round bur (#BR-45) under copious water spray

Isolation: Rubber dam

Procedure:

Pre-operative Steps:

Informed consent obtained

Patient assessment: history, clinical examination, vitality testing, radiographs

Operative Steps:

Group I (Biodentine):

Caries removed and cavity prepared

Biodentine mixed per manufacturer's instructions and placed

After 1 week, a GIC base applied

Final composite restoration placed

Post-op radiograph taken

Group II (Calcium Hydroxide):

Caries removed and cavity dried

0.5 mm Dycal applied and allowed to set (2-3 min)

GIC base placed immediately afterward

Final composite restoration after 1 week

Post-op radiograph taken

Follow-Up Intervals:

2 weeks

6 weeks

12 weeks

Evaluation Criteria:

Clinical Parameters:

Pain (reversible or persistent)

Tenderness to percussion

Response to pulp vitality tests

Radiographic Parameters:

Presence or absence of periapical radiolucency

Periodontal ligament (PDL) space widening

Data Collection Tool:

Data was recorded using a structured proforma (Annexure-C), documenting all clinical and radiographic parameters at baseline and follow-up intervals.

Statistical Analysis:

Software: SPSS Version 26

Quantitative Variables: Mean ± standard deviation (e.g., age, weight)

Qualitative Variables: Frequency and percentage (e.g., pain, radiographic changes)

Test Used: Chi-square test

Level of Significance: p < 0.05 considered statistically significant

Ethical Considerations:

Approved by Institutional Review Board (IRB) and College Ethical Committee

Written informed consent obtained in both English and Urdu

Patient confidentiality strictly maintained

Participants allowed to withdraw at any time without affecting treatment

Budget and Funding:

Funded by Dental College, HITEC-IMS, Taxila

No financial burden on participants

Estimated duration for study completion: 1 year

Expected Outcome:

The study aims to determine whether Biodentine, with its superior physical and biological properties, provides better clinical and radiographic outcomes in indirect pulp capping procedures compared to Calcium Hydroxide in mature permanent teeth.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in the study:

* Age: 20 to 45 years.
* Tooth Type: Mature permanent teeth (maxillary or mandibular).
* Caries Status: Occlusal carious lesions without previous restorations.
* Pulpal Diagnosis: Reversible pulpitis confirmed by:
* Patient history and clinical examination
* Positive response to thermal (cold) and electric pulp tests
* No tenderness to percussion
* Radiographic Assessment: Carious lesion corresponding to ICDAS radiographic score RC-5.
* Periapical Status: No signs of periapical radiolucency or root resorption on radiograph.

Exclusion Criteria:

* Participants will be excluded if they meet any of the following:
* Teeth exhibiting signs of irreversible pulpitis or pulp necrosis.
* Tenderness to percussion on clinical examination.
* Pulp exposure during caries removal.
* Systemic conditions that may interfere with healing or immune response, including:

Chronic systemic illness

Immunocompromised status

Pregnancy

-Third molars (due to anatomical and treatment variability)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Radiographic assessment by Periapical Index (PAI) | Follow-up Timeline for Each Patient: Patients will be evaluated at the following intervals after the indirect pulp capping procedure: Baseline (Initial Treatment) 2 weeks follow-up 6 weeks follow-up 12 weeks follow-up
  PAI Scoring Criteria:
  Score Radiographic Features Interpretation
  1. Normal periapical structures Healthy PDL and periapical tissues
  2. Small changes in bone structure (slight PDL widening) Mild changes; potentially reversible
  3. Changes in bone structure with mineral loss Moderate periapical inflammation
  4. Well-defined radiolucent area Established periapical periodontitis
  5. Severe radiolucency with bone destruction Advanced periapical disease
  Application in my Study:
  At each follow-up (2, 6, 12 weeks), periapical radiographs should be:
  Evaluated using the PAI score
  Compared to baseline radiographs
  Scores ≤2 are generally considered favorable outcomes
  Scores ≥3 indicate disease or failure
Visual Analog Scale (VAS) for Pain Measurement | Patients pain level can be measured on the scale at: Baseline 2-week 6-week 12-week follow-up visits
  1. Pain Assessment
  Type: Spontaneous or provoked
  Tool: Patient history and Visual Analog Scale (VAS) for Pain Measurement
  Classification:
  No pain
  Mild/transient pain (indicative of successful pulp healing)
  Moderate to severe pain (suggestive of pulpal inflammation or failure)
  Interpretation:
  Absence of pain considered a positive outcome.
  Persistent or worsening pain may indicate treatment failure or progression to irreversible pulpitis
  Visual Analog Scale (VAS) for Pain Measurement
  Description:
  A 10 cm horizontal line representing a continuum of pain intensity.
  One end (0 cm) represents "No pain", and the other end (10 cm) represents "Worst possible pain".
  Scoring Criteria:
  VAS Score (cm) Pain Intensity 0 No pain 1-3 Mild pain 4-6 Moderate pain 7-10 Severe pain
  Application in my Study: Patients can be asked to mark their pain level on the scale at:
  Baseline
  2-week
  6-week
  12-week follow-up visits
Tenderness to Percussion | Patients tenderness to percussion will be checked at: Baseline 2-week 6-week 12-week follow-up visits
  2. Tenderness to Percussion
  Tool: Blunt end of dental mirror gently tapped on the occlusal surface
  Response Categories:
  Absent: No discomfort or pain on percussion (favorable response)
  Present: Pain on percussion, indicating potential periapical inflammation or pulp degeneration
  Interpretation:
  Lack of tenderness is a favorable clinical outcome.
  Positive percussion response may suggest underlying periapical involvement or pulpal pathology.
Pulp Vitality Testing : Cold test (Endo-Ice or refrigerant spray on cotton pellet) and Electric Pulp Test (EPT) | Patients tooth vitality testing will be done at: Baseline 2-week 6-week 12-week follow-up visit
  Pulp Vitality Testing
  Methods Used:
  Cold test (Endo-Ice or refrigerant spray on cotton pellet)
  Electric Pulp Test (EPT)
  Response Categories:
  Normal response: Short, sharp, non-lingering sensation (indicative of vital pulp)
  Exaggerated or lingering pain: Suggestive of reversible/irreversible pulpitis
  No response: Indicative of non-vital or necrotic pulp
  Interpretation:
  A normal response to cold or EPT at follow-up implies successful preservation of pulp vitality.
  No response or lingering pain may indicate pulp necrosis or treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Dr Zahoor Dr Zahoor khan, BDS, FCPS, Principal Investigator — Dental college HITEC-IMS Taxila; Dr Zahoor khan, Principal Investigator — Dental college HITEC-IMS Taxila
Locations (1):
- HITEC-IMS Taxila, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: In above URL section the related article link has been provided just for reference & support of study as my study has not been published yet — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5364749/